CLINICAL TRIAL: NCT00264680
Title: Validation Of Qolie-10 For Epilepsy, Comparison Of Quality Of Life In Patients Treated With Lamotrigine Or Valproic Acid
Brief Title: Spanish Validation Of Quality of Life Questionnaire (QOLIE-10) For Epilepsy
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: LAM-2003-01
Record Dates: First submitted 2005-12-09; First posted 2005-12-13 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Epilepsy
Keywords: quality of life; qolie-10; epilepsy; lamotrigine; Validation of questionnaire
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: lamotrigine
Drug: valproic acid
  Other Names: lamotrigine

SUMMARY:
Validation of qolie-10, an epilepsy specific quality of life questionnaire in patients treated with lamotrigine or valproic acid. Comparison of quality of life of epileptic patients treated with lamotrigine or valproic acid. Determination and assessment of the comparative safety of lamotrigine or valproic acid. Assessment and comparison of body image perception in women treated with lamotrigine or valproic acid.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of epilepsy and normal neurological examination.
* Patients receiving lamotrigine or valproic acid at stable doses in monotherapy initiated 2 -4 months before.

Exclusion criteria:

* Pregnant or lactating women.
* Previous treatment with lamotrigine or valproic acid.
* Secondary epilepsy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 333 (Actual)
Dates: Start 2003-10-01 (Actual); Primary Completion 2006-03-01 (Actual); Study Completion 2006-03-01 (Actual)

PRIMARY OUTCOMES:
1. Validity, feasibility and reliability of qolie-10 (test-retest, internal consistency) 2. Qolie-10 scores between groups 3. Body image scores between groups

SECONDARY OUTCOMES:
Adverse Events: nature and number between groups

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline